CLINICAL TRIAL: NCT00126763
Title: An Open-Label, Long-Term Safety Study to Evaluate the Safety of the ZR-02-01 Matrix Transdermal Fentanyl Patch for the Treatment of Moderate to Severe Non-Malignant Chronic Pain
Brief Title: Fentanyl Transdermal Matrix Patch ZR-02-01 to Treat Chronic, Moderate to Severe Non-Malignant Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PK results suggested product did not meet requirement for further development.
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZMF-303
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: Chronic Pain; Pain
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Matrix Transdermal Fentanyl Patch (Experimental)
  Interventions: Drug: Fentanyl Transdermal Matrix Patch ZR-02-01

INTERVENTIONS:
Drug: Fentanyl Transdermal Matrix Patch ZR-02-01 — ZR-02-01 patch contains fentanyl dispersed in a solid matrix, and was available in 25, 50,75 and 100 mcg/hr patches. For patients who were using transdermal fentanyl (ie,Duragesic®), the initial dose of ZR-02-01 was the same as their current Duragesic dose. For patients who were taking oral opioids, the initial dose of ZR-02-01 was determined by the investigator using sponsor-provided conversion guidelines. The patches were worn on the chest or upper arm and an overlay was placed over the patch. Patches (and overlays) were replaced every 3 days
  Other Names: ZR-02-01

SUMMARY:
The purpose of this study is to evaluate the safety of the matrix fentanyl patch ZR-02-01 in providing relief of non-malignant chronic pain.

DETAILED DESCRIPTION:
This study will evaluate the safety of the matrix fentanyl patch. The study will be conducted in opioid-tolerant patients with moderate to severe non-malignant chronic pain currently taking an around-the-clock opioid. Patients will discontinue their current opioid regimen and begin using ZR-02-01 as soon as possible under the direction of the physician investigator upon entry into the study. Patient's dose of ZR 02 01 will be determined by the investigator using sponsor-provided conversion. Pain therapy will be under the supervision of the physician investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 and no older than 75 years of age
* Patient has moderate to severe, non-malignant chronic pain that is expected to last for at least 12 months and is currently taking an around-the-clock opioid to treat his/her pain
* Patient is already receiving opioid therapy, has demonstrated opioid tolerance, and requires a total daily dose of opioids at least equivalent to 25 mcg/hr of transdermal fentanyl. Patients who are considered opioid-tolerant are those who have been taking a daily dose of at least 30 mg of oral morphine or morphine equivalent opioid for at least 2 weeks.

Exclusion Criteria:

* Patient has active cancer
* Patient has a history of substance abuse or has a substance abuse disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse eventsTo | 12 months
  Evaluate the safety of long-term administration of the ZR-02-01 patch for the treatment of moderate to severe, non-malignant chronic pain

SECONDARY OUTCOMES:
Pain Intensity | 12 months
  Patient will rate pain intensity using a 100 mm VAS in which "0" equals "No Pain" and "100" equals "The Worst Pain You Can Imagine." Patients will be instructed on how to use the VAS and will base their response on the average pain that they experienced over the previous 24 hours. VAS will be collected at all study visits except screening.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rauck, MD, Principal Investigator — The Center for Clinical Research
Locations (6):
- United States (6):
  - Arizona Reserach Center, Phoenix, Arizona
  - Loma Linda Center for Pain Management, Loma Linda, California
  - Drug Studies America, Marietta, Georgia
  - Pain Management Institute, Overland Park, Kansas
  - Pain Management Associates, Kansas City, Missouri
  - The Center for Clinical Research, Winston-Salem, North Carolina